CLINICAL TRIAL: NCT05289310
Title: Effects of Daily Low Oxygen Exposure on Weight Status, Body Composition, and Metabolic Health
Brief Title: Low Oxygen Exposure and Weight Status
Acronym: LOWS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Claire Berryman, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBRC 2022-046; 1R01DK127162-01A1 (NIH)
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Body weight; Normobaric hypoxia; Negative energy balance; Energy intake; Energy expenditure
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric hypoxia (NH) (Experimental): 8 weeks of overnight exposure (8 hrs/night) to NH conditions (~15% oxygen; achieved with nitrogen dilution, equivalent to ~8500 feet elevation) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Other: Normobaric hypoxia (NH)
- Normobaric normoxia (NN) (Sham Comparator): 8 weeks of overnight exposure (8 hrs/night) to NN conditions (~21% oxygen; sea level) using a commercially available tent and generator system (Hypoxico, Inc., New York, NY).
  Interventions: Other: Normobaric normoxia (NN)

INTERVENTIONS:
Other: Normobaric hypoxia (NH) — Low oxygen exposure to mimic ~8500 feet elevation (experimental).
  Arms: Normobaric hypoxia (NH)
Other: Normobaric normoxia (NN) — Normal oxygen exposure to mimic sea level conditions (sham comparator).
  Arms: Normobaric normoxia (NN)

SUMMARY:
The objective of the proposed double-blind, parallel-arm, randomized clinical trial is to evaluate changes in body weight and composition, assess determinants of energy balance (intake and expenditure), and measure modulators of energy balance, following 8 wk of calorie restriction (-500 kcal/d) in combination with either overnight exposure to normobaric hypoxia (8 h/night, 15% FiO2, ~2640 m) or normoxia (8 h/night, 21% FiO2), using a commercially available, in-home tent system, in adults with obesity.

DETAILED DESCRIPTION:
Obesity and associated metabolic conditions are a significant public health burden, costing the U.S. ~$150 billion annually. Obesity is both a disease, affecting 1 in 3 Americans, and a risk factor for other chronic diseases, such as cardiovascular disease, type 2 diabetes, and 13 forms of cancers. Diet and exercise are the cornerstone of obesity prevention and treatment. However, a considerable number of individuals are non-responsive to existing weight-loss interventions and obesity rates continue to rise. Therefore, non-conventional approaches are needed to supplement current weight-loss strategies. Daily exposure to low-oxygen conditions may aid in current weight- loss strategies. Moderate (1500-3500 m) and higher (≥ 3500 m) altitude environments are naturally hypoxic due to the lower atmospheric pressure (for reference, Denver, CO is ~1600 m and Mt. Hood in Oregon is ~3500 m). Studies show that sea-level natives exposed to moderate- or high- altitude continuously for 5 or more days lose weight, which is a consequence of prolonged reductions in blood and tissue oxygenation that lead to increased energy expenditure and decreased appetite. However, implementation of hypoxia as a means for weight loss has been limited, to date, by the logistical constraints of traveling to remote locations or access to an altitude chamber. A safe, less expensive, and more logistically feasible alternative is the use of commercially available, low-oxygen systems at sea level, which create a normobaric hypoxic environment. Whether in-home, overnight, normobaric hypoxic exposure, compared to normobaric normoxic exposure, promotes body mass loss in adults with obesity remains unknown. Furthermore, determinants of energy balance, including energy intake and expenditure, and their relative contribution to normobaric hypoxia-induced weight loss have not been investigated. The objective of the proposed double-blind, parallel-arm, randomized clinical trial is to evaluate changes in body weight and composition, assess determinants of energy balance (intake and expenditure), and measure modulators of energy balance, following 8 wk of calorie restriction (-500 kcal/d) in combination with either overnight exposure to normobaric hypoxia (8 h/night, 15% FiO2, ~2640 m) or normoxia (8 h/night, 21% FiO2), using a commercially available, in-home tent system, in adults with obesity. Chronic (8 weeks), overnight (8 hours/night) low oxygen exposure may provide a non-conventional approach to supplement current weight-loss strategies, inform new strategies to accelerate weight loss, aid long-term weight management efforts, and benefit metabolic health in individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI between 30-39.9 kg/m2)
* Born at altitudes below 2,100 meters (~7,000 feet)
* Currently residing in Tallahassee, Florida or surrounding area
* Completed a full FDA authorized or approved COVID-19 vaccination series at least 14 days before any in-person human research activity.
* Not taking any medication(s) that interfere with oxygen delivery/transport for 4 weeks prior to and throughout the entire study (e.g., includes sedatives, sleeping aids, tranquilizers and/or any medication that depresses ventilation, diuretics, alpha and beta blockers).
* Willing to refrain from smoking, vaping, chewing tobacco, and dietary supplement use throughout the entire study.
* Willing to have a hypoxic tent set-up in their home and spend 8 consecutive hours per night in the tent for 8 weeks
* Lives with a family member, partner/spouse, or roommate who can hear and respond in the unlikely event that the blood oxygen, air oxygen, or air carbon dioxide monitoring alarm would sound.

Exclusion Criteria:

* Living in areas that are more than 1,200 m (~4,000 feet), or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months
* Individuals who have not completed a full FDA authorized or approved COVID-19 vaccination series at least 14 days before any in-person human research activity.
* Cardiovascular abnormalities, gastrointestinal disorders, or any condition that interferes with oxygen delivery/transport (e.g., kidney disease, cardiovascular disease, etc.)
* Oxygen saturation < 95% while awake or oxygen saturation dips below 88% for a total of ≥ 10 min overnight in normoxic conditions
* Evidence of apnea or other sleeping disorders
* Evidence of prior high-altitude pulmonary edema (HAPE) or high-altitude cerebral edema (HACE) diagnosis
* Diagnosis or family history of sickle cell anemia/trait
* Hematocrit <42% for males, <36% for females
* Hemoglobin <13 g/dL for males, <12 g/dL for females
* Blood donation within 8 weeks of beginning the study
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Women who are pregnant, lactating, planning to become pregnant, or who have had an irregular menstrual cycle in the past 6 mo.
* Weight gain or loss > 10% of body weight during the past 6 months
* Adults unable to consent

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 10 weeks (70 days)
  Body weight will be measured during the baseline weight maintenance phase (days -14 to 0) and each morning during the study (days 1 to 56) following an overnight fast and morning void, using a calibrated digital scale provided to participants to use at home (A&D Medical wireless weight scale UC-352BLE, San Jose, CA). Change in body weight will be calculated as: body weight on day 56 - baseline body weight (average of days -14 to 0).

SECONDARY OUTCOMES:
4-compartment body composition using DEXA and deuterium dilution | Days -7 and 49
  Body composition will be determined following at least a 10 hour fast and morning void on day -7 and 49 using dual energy x-ray absorptiometry (DEXA, Discovery W, Hologic Inc., Bedford, MA or equivalent). The volunteer will remove all metal-containing objects from their body, lay face-up on the DEXA densitometer table in light clothing (t-shirt, shorts, socks), and be asked to remain motionless for the 8-10 min scan. A scanner emitting low energy x-rays and a detector will pass over the participant. These data will be used to calculate total body mass, fat-free mass, fat mass, and bone mass. Total body water will be measured following at least a 10 hour fast and 1 hour without water intake using oxygen-18 labeled water on days -7 and 49.
Waist circumference | Days -7 and 49
  Waist circumference will be measured to the nearest centimeter using a measuring tape. Measurements will be taken in duplicate.
Blood volume | Days -7 and 49
  Blood volume will be determined using the optimized carbon monoxide rebreathing method on days -7 and 49. In this method, a finger stick blood sample is taken and basal carboxyhemoglobin concentrations determined using a blood gas analyzer (OSM-3, Radiometer). Carbon monoxide is then inhaled via a spirometer (SpiCo, Blood Tec.) for 2 min. Seven minutes after inhaling the carbon monoxide bolus, a second finger prick blood sample is taken to determine the increase in carboxyhemoglobin concentration. The change in percentage of carboxyhemoglobin between the basal and second measurements can be used to calculate hemoglobin mass and blood volume.
Total daily energy expenditure (TDEE) | Days -7 to 0 and 49-56
  Energy expenditure will be assessed by the doubly labeled water (DLW) method. Briefly, upon waking, volunteers will provide a urine sample and completely void their bladder, this sample will be used to measure background isotope enrichment. The participant will then consume 1.5 g/kg of 10% O18 and 0.06 g/kg of deuterium. Urine samples will be collected at 4 h, 6.5 h, 24 h, 3 d, 5 d, and 7 d after dosing.
Resting metabolic rate | Days 0 and 56
  Resting metabolic rate will be measured with open circuit, indirect calorimetry (ParvoMedics TrueOne 2400 metabolic cart, Sandy, UT) in the morning, upon arrival to the lab on days 0 and 56.
Resting substrate oxidation | Days 0 and 56
  Resting substrate oxidation will be measured with open circuit, indirect calorimetry (ParvoMedics TrueOne 2400 metabolic cart, Sandy, UT) in the morning, upon arrival to the lab on days 0 and 56.
Ad libitum energy intake | Days 0 and 56
  Participants will be provided an ad libitum mixed-macronutrient meal (e.g., frozen lasagna) on days 0 and 56. Food will be provided in excess of expected consumption for one individual. Water in the amount of 240 g will be provided during the meal. Participants will be instructed to consume all water before completing the meal and will not be permitted additional water during the meal, in order to control the effect of fluid intake on satiety. To limit social influence on eating behavior, each ad libitum meal will be consumed in isolation. Leftover food will be collected and weighed after participants have left the laboratory. Energy and nutrient content of the amount consumed will be determined using Food Processor software (version 11.6.0, ESHA Research, Salem, OR) under the supervision of a Registered Dietitian.
Subjective appetite measures | Days 0 and 56
  Subjective appetite will be measured on study days 0 and 56. Subjectively rated appetite will be assessed immediately before the oral glucose tolerance test (OGTT), at 15, 30, 45, 60, 90, and 120 minutes after beginning the OGTT, and upon cessation of the ad libitum meal (discussed above) using 100 mm visual analog scales to rate fullness, hunger, desire to eat, and prospective food consumption. Composite satiety score will be calculated from the individual appetite scores using the equation: CSS = (fullness + (100 - Desire to eat) + (100 - Hunger) + (100 - Prospective food consumption) / 4.
Overnight oxygen saturation (wrist-worn device) | 10 weeks (70 days)
  Participants will be provided a wrist-worn device with Bluetooth capabilities (vivosmart 4, Garmin, Olathe, KS) to be worn for 2 weeks prior to the start of the study (baseline measurement) and continuously for the entirety of the study. This devise will measure steps, physical activity levels, heart rate, overnight oxygen saturation, and sleep patterns.
Overnight oxygen saturation (index finger pulse oximetry) | 10 weeks (70 days)
  In addition to the wrist-worn physical activity monitoring device (vivosmart 4, Garmin, Olathe, KS) that will measure overnight oxygen saturation, participants also will wear a pulse oximeter (PalmSAT® 2500A) on their index finger overnight to measure oxygen saturation.
Prevalence of acute mountain sickness | Days 0-7, 14, 21, 28, 35, 42, and 56
  The prevalence and severity of AMS will be determined from information gathered using the shortened version of the Environmental Symptoms Questionnaire (ESQ) and the Lake Louise AMS Scoring System (LLS; 5 min; 26 questions total). At completion of the questionnaire, oxygen saturation will be determined using finger pulse oximetry (PalmSAT® 2500A, Nonin Medical, Inc., Plymouth, MN). AMS and oxygen saturation measurements will be taken in the morning (between 5:00-8:00am, inside tent) and evening (9:00pm-12:00am, inside tent) on days 0-7, 14, 21, 28, 35, 42, and 56.
Heart rate variability | Days 0 and 56
  A 3-lead electrocardiogram will be conducted on days 0 and 56 to assess heart rate variability. Participants will have electrode patches placed on their chest to measure the electrical activity of the heart.
Heart rate variability | 10 weeks (70 days)
  Participants will be provided a wrist-worn device with Bluetooth capabilities (vivosmart 4, Garmin, Olathe, KS) to be worn for 2 weeks prior to the start of the study (baseline measurement) and continuously for the entirety of the study. This devise will measure steps, physical activity levels, heart rate, overnight oxygen saturation, and sleep patterns.
Urinary epinephrine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Epinephrine concentrations in the urine samples will be measured.
Urinary norepinephrine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Norepinephrine concentrations in the urine samples will be measured.
Urinary dopamine | Days -1, 13, and 55
  On days -1, 13, and 55 urine will be collected during the overnight time period. Participants will void their bladder before entering the tent in the evening (they will not collect this portion). Participants will collect any urine produced throughout the night and will collect one final time in the morning after exiting the tent. Dopamine concentrations in the urine samples will be measured.
Plasma glucose concentrations | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Plasma insulin concentrations | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Whole-body insulin sensitivity index | Days 0 and 56
  A 75-g oral glucose tolerance test (OGTT) will be conducted on days 0 and 56. A venous catheter will be placed and blood samples obtained at -5, 30, 60, 90, and 120 min during the OGTT for measurements of plasma glucose and insulin concentration. Insulin sensitivity will be determined by using the whole-body insulin sensitivity index (WBISI), also known as the Matsuda Index.
Thermic effect of glucose | Days 0 and 56
  The thermic effect of glucose will be measured on study days 0 and 56 with open circuit, indirect calorimetry (2400 TrueOne, Parvo Medics) using established protocols. Resting metabolic rate measurements will be taken prior to glucose administration in a thermo-neutral room while the participant is in the supine position (as described above). During the oral glucose tolerance test the thermic effect of glucose will be measured in 15 min increments for 2 hours (15-30, 45-60, 75-90, and 105-120 minutes).
24-hour continuous glucose concentrations | Days -14-0, 1-14, and 42-56
  A continuous glucose monitor (Freestyle Libre Pro) will be inserted into the subcutaneous adipose tissue behind the arm and will be used to collect and assess 24-hour glucose concentrations.
24-hour glucose variability | Days -14-0, 1-14, and 42-56
  A continuous glucose monitor (Freestyle Libre Pro) will be inserted into the subcutaneous adipose tissue behind the arm and will be used to collect and assess 24-hour glucose concentrations.
Assessment of sleep | 10 weeks (70 days)
  Participants will be provided a wrist-worn device with Bluetooth capabilities (vivosmart 4, Garmin, Olathe, KS) to be worn for 2 weeks prior to the start of the study (baseline measurement) and continuously for the entirety of the study. This devise will measure steps, physical activity levels, heart rate, overnight oxygen saturation, and sleep patterns.
Pittsburgh Sleep Quality Index | Days -1, 14, and 56
  The Pittsburgh Sleep Quality Index will be used to examine participant sleep quality on days -1, 14, and 56 (5 min; 18 questions total).
Subjective sleep quality | Days -7-0, 1-14, and 49-56
  Participants will be asked to complete a sleep diary before and after sleep for 7 d at baseline, on days 0-14, and on days 49-56. The sleep diary includes questions related to mood, caffeine intake, substance use (e.g. alcohol, caffeine, and prescriptions), and sleep quality.
Fasting measures of iron status | Days 0 and 56
  Serum iron, total iron binding capacity, soluble transferrin receptor, hepcidin, hemoglobin, hematocrit, ferritin, erythroferrone, and erythropoietin will be measured in fasting blood samples collected on days 0 and 56.
Psychosocial Factors | Days 0, 14, and 56
  The Positive and Negative Affect Schedule (PANAS), Cohen Perceived Stress Scale, Big Five Inventory-2, Delay Discounting questionnaire, Palatable Eating Motives Scale, and the Generalized Self-Efficacy scale will be administered on day 0, 14, and 56.
Fasting blood pressure | Days -7 and 49
  Participants will rest in a seated position for at least 5 minutes before an automated blood pressure cuff is used to measure blood pressure in triplicate.
Barrier Questionnaire | Day 56
  This questionnaire will be administered to participants on day 56 to assess real and perceived barriers to sleeping in a hypoxic tent (5 min; 17 questions total).
Change in body weight | 4 weeks after intervention ends
  Body weight also will be measured 4 weeks after the study intervention ends to assess whether weight loss is sustained. Change in body weight will be calculated as:
  * Body weight on day 84 (i.e., 4 wk post-intervention) - baseline body weight (average of days -14 to 0)
  * Body weight on day 84 (i.e., 4 wk post-intervention) - body weight on day 56

CONTACTS AND LOCATIONS:
Overall Officials: Claire E. Berryman, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riley TM, Weschenfelder C, Ravussin E, Rood JC, Greenway F, Taff S, Hickner RC, Cao H, Sutin AR, Todd G, Hennigar SR, Berryman CE. Effects of daily low oxygen exposure on weight status, body composition, and metabolic health in adults with obesity: protocol for a randomized, double-blind, controlled-feeding study. Contemp Clin Trials. 2026 Jan;160:108167. doi: 10.1016/j.cct.2025.108167. Epub 2025 Nov 26. PMID 41314599